CLINICAL TRIAL: NCT06846632
Title: Graftless Technique in Open Maxillary Sinus Lifting Using Poly-Ether-Ether-Ketone Versus Titanium Meshwork for Evaluation of Bone Quantity: Randomized Clinical Trials
Brief Title: Graftless Technique in Open Maxillary Sinus Lifting Using PEEK Versus Ti -Meshwork
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, mohamed gamal hammad, MSc degree of oral and maxillofacial surgery, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 33-6-24
Record Dates: First submitted 2025-02-16; First posted 2025-02-26 (Actual); Last update posted 2025-02-26 (Actual); Status verified 2025-02

CONDITIONS: Maxillary Sinus
Keywords: maxillary sinus lifting , PEEK , titanium meshwork

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- placement of titanium meshwork after maxillary sinus lifting (Experimental): placement of titanium meshwork after maxillary sinus lifting
  Interventions: Device: titanium meshwork
- placement of PEEK after maxillary sinus lifting (Experimental): placement of PEEK after maxillary sinus lifting
  Interventions: Device: PEEK

INTERVENTIONS:
Device: PEEK — placement of PEEK after maxillary sinus lifting
  Other Names: poly ether ether ketone
  Arms: placement of PEEK after maxillary sinus lifting
Device: titanium meshwork — placement of titanium meshwork after maxillary sinus lifting
  Arms: placement of titanium meshwork after maxillary sinus lifting

SUMMARY:
The aim of the study is to assess the amount of bone formation with PEEK (intervention group) in comparison with Titanium Meshwork (control group) in maxillary sinus lifting using CBCT and assessment of the biocompatibility of the Meshwork and PEEK with the schniederian membrane integrity.

DETAILED DESCRIPTION:
All patients involved in this study will be divided into two equal groups, each group will be; (Tested group): PEEK after maxillary sinus lifts (Caldwell luc approach). (Control group): Titanium meshwork after maxillary sinus lifts (Caldwell luc approach).

Clinical evaluation:

A through medical and dental history followed by clinical examination was carried out for all patients. Clinical measurements were taken to ensure patient adherence to our initial inclusion criteria prior to further investigations.

A preoperative digital panoramic radiograph with 1:1 magnification was taken for each patient as a primary survey in order to exclude the presence of any lesion at the area of interest and take a primary measurement for the residual bone height of maxillary sinus.

CBCT will be taken in order to design the custom-made PEEK model and its guide of external window before the milling.

Intra operative procedures for two groups:

The operation was carried out with the patient under local anesthesia (2% Lido HCl with 1:100,000 epinephrine). The perioral areas were aseptically prepared. A crestal incision was made on the midline of the gingiva attached to the edentulous ridge. The flap was elevated carefully and extended labially to expose the bone. A mesial and distal vertical releasing incision will be made as needed. The mucosal flap was denuded subperiosteally to fully expose the sharp and thin alveolar ridge and the lateral wall of the maxillary sinus. Extreme care was taken to radically elevate the sinus membrane from the lateral access window opened by using an electric-motor drill with appropriate water cooling. The floor, lateral wall, medial and posterior wall of the sinus membrane were meticulously detached and pushed upward for the placement of PEEK in intervention group and titanium meshwork in control group.

• Follow up: Patients will be evaluated after 3 days and weekly for the first month and then after 6 months Radiographic assessment will be achieved by CBCT scan 6 months postoperatively to calculate the amount of vertical bone gain.

ELIGIBILITY:
Inclusion Criteria:

* • Posterior edentulous ridges with pneumatized maxillary sinus and remaining bone height of 3 to 6 mm.

  * Patient age ranges from 25 to 50 years.
  * ASA physical status I and II.
  * Patients willing to be a part of the study and ready to give their consent in writing for the same.
  * Patient not complains from maxillary sinusitis
  * Patients are free from T.M.J disorders, abnormal oral habits such as bruxism.
  * Patient with good oral hygiene.

Exclusion Criteria:

* • Untreated gingivitis, periodontitis.

  * Subjected to irradiation in the head and neck area less than 1 year before implantation.
  * Untreated periodontitis.
  * Insufficient oral hygiene and motivation.
  * Pregnant or nursing.
  * Bone pathology.
  * Patient with blood disease.
  * Patient with any systematic disease that may affect normal healing.
  * Active infection or severe inflammation in the area intended for implant placement.
  * Treated or under treatment with intravenous amino-bisphosphonates.

Ages: 25 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2024-05-03 (Actual); Primary Completion 2024-10-03 (Actual); Study Completion 2024-11-03 (Actual)

PRIMARY OUTCOMES:
Bone quantity | at 6 months of maxillary sinus lifting
  assessment of bone quantity using CBCT

SECONDARY OUTCOMES:
Compatibility with Schneiderian membrane | at 6 months of maxillary sinus lifting
  assessment of the biocompatibility with Schneiderian membrane

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Dentistry Cairo University, Cairo, Egypt